CLINICAL TRIAL: NCT06483425
Title: A Biomarker Exploration Study of Precision Treatment in Ovarian Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Qinglei Gao, Professor, Tongji Hospital
Other Study IDs: 2024-TJ-OCBiomarker
Record Dates: First submitted 2024-06-24; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Ovarian Cancer; Biomarker
MeSH Terms: conditions — Ovarian Neoplasms | interventions — RNA; Proteins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Tumor, Ascite, and other samples would be collected for sequencing for the identification of biomarkers for OC treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ovarian cancer pateitns: Patients diagnosed with Ovarian cancer in Tongji Hospital, Wuhan.
  Interventions: Genetic: Sequencing of DNA, RNA, and Proteins

INTERVENTIONS:
Genetic: Sequencing of DNA, RNA, and Proteins — Sequencing of DNA, RNA, and Proteins for Tumor, Blood, Ascite, and other samples before and after treatment.

SUMMARY:
This clinical trial aims to investigate the role of biomarkers in guiding precision treatment for ovarian cancer. The study will explore the effectiveness of personalized treatment strategies based on specific biomarkers identified in ovarian cancer patients. By analyzing the correlation between biomarker profiles and treatment outcomes, the trial seeks to optimize treatment decisions and improve overall survival rates in ovarian cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with ovarian cancer.
* Willingness to undergo biomarker testing.
* Ability to provide informed consent for participation in the study.

Exclusion Criteria:

* Inability to comply with study requirements or follow-up visits.
* Previous participation in a conflicting clinical trial.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Ovarian cancer patients.
Study Population: Patients diagnosed with Ovarian cancer, who are willing to participate in this study and agree to donate samples for sequencing could be included.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Biomarker explorarion | 5 years
  Blood, tumor, and other samples should be sequenced by RNA-seq, Next-Generation Sequencing, or proteomics to identify specific biomarkers associated with treatment response and prognosis in ovarian cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No